CLINICAL TRIAL: NCT03041051
Title: Study of the Immunogenicity and Immunological Memory Induced by the 13valent Pneumococcal Conjugate(PCV13) and 23valent Plain Polysaccharide Vaccine(PPV23) in HIV-infected Adults
Brief Title: Immunological Memory Induced by the 13valent Pneumococcal Conjugate(PCV13) and 23valent Plain Polysaccharide Vaccine(PPV23) in HIV-infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Principal Investigator, Vana Spoulou, Associate Professor of Pediatric Infectious Diseases, Aghia Sophia Children's Hospital of Athens
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 51198eAS
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCV13 (Experimental)
  Interventions: Biological: PCV13
- PPV23 (Experimental)
  Interventions: Biological: PPV23

INTERVENTIONS:
Biological: PCV13
  Arms: PCV13
Biological: PPV23
  Arms: PPV23

SUMMARY:
The purpose of this study is to determine the effect of a combined vaccination schedule of the 13-valent pneumococcal conjugate (PCV13) and 23valent plain polysaccharide vaccine (PPV23) on the establishment of immunological memory in HIV-infected adults on ART.

ELIGIBILITY:
Inclusion Criteria:

* CD4 T cell count >200cells/μl
* on ART

Exclusion Criteria:

* no previously recorded allergy to PCV, PPV23
* no intravenous immunoglobulin (IVIG) given within the previous 6 months
* no other vaccine given within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
immunoglobulin G (IgG) B memory cell response one month post vaccination (measured by flow cytometry) | One month post-PCV13, PPV23
  immunoglobulin G (IgG) B memory cell response one month post vaccination (measured by flow cytometry)
immunoglobulin M (IgM) B memory cell response one month post vaccination (measured by flow cytometry) | One month post-PCV13, PPV23
  immunoglobulin M (IgM) B memory cell response one month post vaccination (measured by flow cytometry)

CONTACTS AND LOCATIONS:
Overall Officials: Vana Spoulou, Principal Investigator — Greece 'Aghia Sophia' Children's Hospital Athens, Attiki, Greece, 11527

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farmaki PF, Chini MC, Mangafas NM, Tzanoudaki MT, Piperi CP, Lazanas MZ, Spoulou VS. Immunogenicity and Immunological Memory Induced by the 13-Valent Pneumococcal Conjugate Followed by the 23-Valent Polysaccharide Vaccine in HIV-Infected Adults. J Infect Dis. 2018 Jun 5;218(1):26-34. doi: 10.1093/infdis/jiy135. PMID 29722823